CLINICAL TRIAL: NCT00301496
Title: Randomized Controlled Eight Week Cross-over Clinical Evaluation of the 3M Coban 2-Layer Compression System to Evaluate the Product Performance in Patients With Venous Leg Ulcers
Brief Title: Randomized Controlled 8-week Crossover Evaluation of Compression Bandage Systems for Venous Leg Ulcers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Solventum US LLC (Industry)
Collaborators: 3M (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 05-010302
Record Dates: First submitted 2006-03-10; First posted 2006-03-13 (Estimated); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Venous Ulcer
MeSH Terms: conditions — Varicose Ulcer

INTERVENTIONS:
Device: Coban 2 Layer Compression System

SUMMARY:
The purpose of this study is to evaluate the product performance of a new 2-layer compression bandage for the treatment of venous leg ulcers.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the product performance of a new 2-layer compression bandage for the treatment of venous leg ulcers. The new bandage is a 2-layer compression system. It will be used over primary dressings to provide the compression that is beneficial to venous leg ulcers.

ELIGIBILITY:
Inclusion Criteria:

* venous leg ulcer
* patient can walk

Exclusion Criteria:

* cancerous ulcers
* diabetic foot ulcer

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80
Dates: Start 2006-03; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Product Performance

CONTACTS AND LOCATIONS:
Overall Officials: Christine Moffatt, PhD, MA, RGN, Principal Investigator — Centre for Research and Implementation of Clinical Practice
Locations (10):
- United States (5):
  - Institute for Advanced Wound Care, Montgomery, Alabama
  - Center for Clinical Research, Inc., Castro Valley, California
  - Gwinnet Hospital System, Lawrenceville, Georgia
  - Wound Healing and Treatment Center - Silver Cross Hospital, Joliet, Illinois
  - Wound Healing Center, Terre Haute, Indiana
- Canada (2):
  - Dermatology Clinic - Montreal General Hospital, Montreal, Quebec
  - Dermatology Clinic, Mississauga, Ontario
- United Kingdom (3):
  - Wound Healing Research Unit, Cardiff
  - Grantham & District Hospital, Grantham
  - Clayponds Hospital, London